CLINICAL TRIAL: NCT00764283
Title: The Prevention of Postoperative Epidural Catheter Migration: a Comparison of Three Types of Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Eric Mortier, University Ghent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008/278
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Tegaderm dressing
  Interventions: Device: Tegaderm dressing
- 2 (Active Comparator): Epi-Fix dressing
  Interventions: Device: Epi-Fix dressing
- 3 (Active Comparator): Lockit-Plus dressing
  Interventions: Device: Lockit-Plus

INTERVENTIONS:
Device: Tegaderm dressing — Tegaderm dressing is used to secure the epidural catheter for postoperative analgesia
  Arms: 1
Device: Epi-Fix dressing — Epi-Fix dressing is used to secure the epidural catheter for postoperative analgesia
  Arms: 2
Device: Lockit-Plus — Lockit-Plus dressing is used to secure the epidural catheter for postoperative analgesia
  Arms: 3

SUMMARY:
Three types of dressing will be compared to prevent postoperative epidural catheter migration. Patients will be randomised to have a Tegaderm dressing, an Epi-fix dressing or a Lockit-Plus dressing to secure the epidural catheter for postoperative analgesia. The length of the epidural catheter visible at the patient's skin surface will be recorded after insertion and every day until removal. The integrity of the dressing and problems with analgesia will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients who receive a lumbar epidural catheter for patient controlled analgesia will be included after informed consent
* 18 years or older

Exclusion Criteria:

* Patients who did not sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Epidural catheter migration from insertion till removal | Until removal of the epidural catheter

SECONDARY OUTCOMES:
Problems of analgesia during Patient Controlled Epidural Analgesia | Until removal of the epidural catheter
Body Mass Index | Until removal of the epidural catheter
The integrity of the dressing | Until removal of the epidural catheter
The comfort of the dressing | Until removal of the epidural catheter

CONTACTS AND LOCATIONS:
Overall Officials: Eric Mortier, MD, PhD, Principal Investigator — University Ghent
Locations (1):
- AZ Maria Middelares Ghent, Ghent, Belgium